CLINICAL TRIAL: NCT01354873
Title: Colorectal Polyp Discrimination Using High-Definition Narrow Band Imaging
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Olympic Medical (Industry)
Responsible Party: Michael B Wallace, MD, Mayo Clinic
Other Study IDs: 10 002315
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Colon Polyps
Keywords: Colonoscopy; Colon Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators seek to compare the accuracy of the existing colonoscope model to determine the magnitude of the improvement the investigators can expect in polyp discrimination as neoplastic or non-neoplastic.

DETAILED DESCRIPTION:
Information will be collected. Images will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Presenting for surveillance, screening or diagnostic colonoscopy
* Willingness to provide informed consent

Exclusion Criteria:

* Inability to provided informed consent
* Pregnancy
* Known inflammatory bowel disease
* Personal or family history of polyposis or nonpolyposis syndrome
* Emergency colonoscopy/endoscopy
* Coagulopathy or thrombocytopenia preventing polypectomy
* Procedure indication for acute bleeding or active colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and Women(not pregnant) presenting to the GI lab for colonoscopy. Child bearing potential not excluded.
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2011-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Accuracy of In Vivo determination of colorectal polyps histopathology | 1 year
  Compare accuracy of current colonoscope to improved colonoscope for discrimination of polyps as neoplastic versus non-neoplastic. The accuracies of the two approaches will be compared via logistic regression model with the significance of the difference in the accuracies assessed via generalized estimating equation approach to take account of the possible dependence introduced by inclusion of mulitple polyps per patient.

SECONDARY OUTCOMES:
Sensitivity and specificity of In Vivo discrimination of colorectal polyp histopathology in white light and narrow band imaging modes. | 1 year
  Estimate the sensitivity and specificity in high definition mode for distinguishing neoplastic from none neoplastic lesions. Sensitivity and specificity will be estimated using the logistic regression approach as above; 95% confidence intervals will be obtained by transforming confidence intervals on the logs odds scale.

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Wallace, MD,MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States